CLINICAL TRIAL: NCT05615350
Title: The Effect of Meal Texture on Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Ciaran Forde, prof.dr. CG (Ciarán) Forde, Wageningen University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: CONSTRUCT
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Eating Behavior
Keywords: Texture; Eating rate; Food intake; Energy intake
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meals served during breakfast (Experimental): Twice a week for six weeks (in total twelve times) participants will consume meals ad libitum during breakfast.
  Interventions: Other: Meals served during breakfast with a wide range of different food textures
- Meals served during lunch (Experimental): Twice a week for six weeks (in total twelve times) participants will consume meals ad libitum during lunch. They will receive a standardized breakfast meal.
  Interventions: Other: Meals served during lunch with a wide range of different food textures

INTERVENTIONS:
Other: Meals served during breakfast with a wide range of different food textures — Ad libitum portions of twelve different meals with a wide range of food textures served during breakfast at the eating behaviour lab
  Arms: Meals served during breakfast
Other: Meals served during lunch with a wide range of different food textures — Ad libitum portions of twelve different meals with a wide range of food textures served during lunch at the eating behaviour lab
  Arms: Meals served during lunch

SUMMARY:
In this study the effect of meal texture differences (slow vs fast eating rate) on intake will be investigated.

DETAILED DESCRIPTION:
Rationale: Food texture modifies eating rate and through that the energy intake of foods. It is shown that harder, chunkier, more viscous, and more voluminous foods decrease eating rate of foods and thus decrease energy intake. However, most research is done in model foods or single foods. So far, little research on food texture and intake has been performed for meals. It is not known what the effect of food texture and eating rate is on intake in a wide variety of meals. Knowledge on the effect of food texture on intake could be used for strategies to drive or limit energy intake.

Objective: The objective is to determine how a wide range of different food textures influence energy intake, food intake, and eating behaviour.

Study design: All participants receive all twelve different meals (within subject design). The meals are either served during breakfast or lunch. The meals have a wide range of different food textures. Participants consume the meals ad libitum twice per week for six weeks long with at least two days in between.

Study population: Healthy Dutch speaking adults (n=30) between 18-55 years old with a BMI between 18.5-30 kg/m2.

Intervention: Participants will join twelve test sessions. For the test sessions they will visit the eating behaviour lab where they receive ad libitum meals during breakfast or lunch. During meal consumption participants are video recorded to determine eating behaviour. The participants will receive in total twelve meals. The order in which participants will receive the meals will be block randomized (block n = 5).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Good appetite
* Between 18 and 55 years old
* Speak and understand English without difficulty
* BMI between 18.5-30 kg/m2.
* Non-smoker
* Commonly (5 out of 7 week days) eat three meals a day every day around the

Exclusion Criteria:

* Have difficulties with swallowing, chewing, and/or eating in general;
* Are suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, respiratory disease, or diabetes
* Have taste or smell disorders
* Have braces or oral piercing (dental wire behind teeth is allowed)
* are smoking
* Consume on average more than 21 glasses of alcohol per week
* Are not willing to stop using drugs during the study period (from inclusion till last test session)
* Use medication that may influence study outcomes
* Have allergies or intolerance to any ingredient of the test meals
* Are not willing to eat the test food because of eating habits, believes, or religion
* Follow a vegetarian or vegan diet
* Are lactose intolerant
* Have facial hair such as a beard
* Follow an energy restricted diet during the last 2 months
* Gained or lost 5 kg of body weight over the last half year
* Are an employee, thesis student or intern at the chair group of Sensory Science and Eating Behaviour Human Nutrition (WUR).
* Do intensive exercising more than 8 hours per week
* Low score (<1) for liking the individual test meals on a nine point Likert scale based on pictures of the meals
* Familiar with at least 75% of the test meals (self-report)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Energy intake (kcal) | 6 weeks
  Energy intake (kcal) of each meal

SECONDARY OUTCOMES:
Food intake (g) | 6 weeks
  Food intake (g) of each meal
Eating rate (g/min) | 6 weeks
  Eating rate (g/min) measured with video recording and automated video analysis

OTHER OUTCOMES:
BMI | 5 minutes
  Obtained by body weight (kg; measured using a weighing scale) and height (cm; measured using a stadiometer) as assessed during screening
Subjective hunger | 6 weeks
  Hunger measured before and after meal consumption on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Subjective fullness | 6 weeks
  Fullness measured before and after meal consumption on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Subjective desire to eat | 6 weeks
  Desire to eat measured before and after meal consumption on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Liking | 6 weeks
  Liking of meals after one bite and after meal consumption will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Flavour intensity | 6 weeks
  Flavour intensity after one bite will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Subjective prospective consumption | 6 weeks
  Prospective consumption measured before and after meal consumption on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Hardness | 6 weeks
  Hardness after one bite will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Thickness | 6 weeks
  Thickness after one bite will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Dryness | 6 weeks
  Dryness after one bite will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Familiarity | 6 weeks
  Familiarity (after one bite and after the meal) will be rated on a 9 point Likert scale
Expected satiation | 6 weeks
  Expected satiation (after one bite) will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Desire to eat the meal | 6 weeks
  Desire to eat the meal (after one bite and after the meal) will be rated on a 100-mm Visual Analogue Scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Reasons for eating cessation | 6 weeks
  Reasons for eating cessation assessed with the Reasons Individuals Stop Eating Questionnaire (RISE-Q)
Self-reported eating rate | 1 minute
  Self-reported eating rate measured using the question "How would you describe your eating rate compared with others?" which can be answered on a five-point Likert scale ('very slow', 'slow', 'average', 'fast' or 'very fast')
Restrained eating, emotional eating and external eating | 30 minutes
  The level of restrained, emotional, and external eating assessed with the Dutch Eating Behaviour Questionnaire (DEBQ) consisting out of 33 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Human Nutrition Department, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No